CLINICAL TRIAL: NCT07339085
Title: Advanced Dual-Nuclei MRI for Differentiation of Recurrent Brain Metastases and Radiation Necrosis
Brief Title: Advanced Magnetic Resonance Imaging for the Identification of Recurrent Brain Tumors and Radiation Necrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-1250; NCI-2025-06605 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-1250 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH); R21CA303383 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Malignant Brain Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aim 1 (advanced MRI) (Experimental): Patients undergo advanced DR-CSI and sodium MRI over 30 minutes prior to SOC surgical resection or biopsy. Patients also undergo clinical MRI and tissue sample collection on study.
  Interventions: Procedure: Advanced Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging
- Aim 2 (advanced MRI) (Experimental): Patients undergo advanced DR-CSI and sodium MRI over 30 minutes before SRS and 2 weeks, 3 months, and 6 months post-SRS. Patients also undergo clinical MRI on study.
  Interventions: Procedure: Advanced Magnetic Resonance Imaging; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Advanced Magnetic Resonance Imaging — Undergo advanced DR-CSI and sodium MRI
  Other Names: AMRI
Procedure: Biospecimen Collection — Undergo tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Aim 1 (advanced MRI)
Procedure: Magnetic Resonance Imaging — Undergo clinical MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This clinical trial studies whether advanced magnetic resonance imaging (MRI) techniques, including diffusion-relaxation correlation spectrum imaging (DR-CSI) and sodium imaging, can be used to identify the difference between brain tumors that come back after a period of improvement (recurrent) and treatment-related tissue damage (radiation necrosis [RN]). Radiation therapy is often used in the treatment of brain tumors. Radiation treatment response can be difficult to assess and is usually done using conventional MRI, which uses radio waves and a powerful magnet linked to a computer to create detailed pictures of areas inside the body. Current imaging techniques have a limited ability to identify the difference between recurrent brain tumor and RN due to their similar appearance on conventional MRI and overlapping clinical presentation. This makes it hard for doctors to plan the best way to treat these tumors. DR-CSI is a new MRI technique with the potential to detect microscopic tissue components with different characteristics. Sodium imaging is an MRI technique that estimates the total sodium concentration in the obtained images. It may be able to identify the small structures within the tissue of brain tumors. Advanced MRI techniques like DR-CSI and sodium imaging may be effective in identifying the difference between recurrent brain tumors and RN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop and validate dual-nuclei microstructural MRI biomarkers to differentiate between recurrent brain metastasis (rBM) and RN.

II. Investigate longitudinal microstructural changes following stereotactic radiosurgery (SRS) treatment and predict clinical outcome.

OUTLINE: Patients are assigned to 1 of 2 aims.

AIM 1: Patients undergo advanced DR-CSI and sodium MRI over 30 minutes prior to standard of care (SOC) surgical resection or biopsy. Patients also undergo clinical MRI and tissue sample collection on study.

AIM 2: Patients undergo advanced DR-CSI and sodium MRI over 30 minutes before SRS and 2 weeks, 3 months, and 6 months post-SRS. Patients also undergo clinical MRI on study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosed with metastatic brain tumor
* AIM 1: Scheduled for surgical resection or tissue biopsy +/- laser interstitial thermal therapy (LITT)
* AIM 2: Scheduled for SRS treatment

Exclusion Criteria:

* Patients with contraindications to MRI, severe renal impairment
* Patients with evidence of disseminated leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Imaging features of recurrent brain metastasis (rBM) and radiation necrosis (RN) (Aim 1) | At time of advanced magnetic resonance imaging: Baseline
  Will compute the diffusion-relaxation (DR) spectra and total sodium concentration (TSC) within biopsy regions of interest and use Student t-test or Mann-Whitney U test, depending on the data distribution, to compare imaging features between rBM and RN groups. Specifically, for DR spectra, the test statistic at each spectral location will be used to identify spectral components associated viable tumor and treatment effect. The information will subsequently be used to partition the voxel-wise DR spectra and compute voxel-wise "viable tumor" and "treatment effect" fraction maps. Multivariate logistic regression models will assess the predictive value of the imaging biomarkers, including DR-correlation spectrum imaging (CSI) spectral components and TSC. Receiver operating characteristic (ROC) analysis will evaluate diagnostic performance, calculating area under the curve, sensitivity, specificity, and optimal cutoff values for differentiating rBM and RN.
Stereotacic imaging-guided biopsies and correlation with tissue quantifications (Aim 1) | Up to completion of surgery
  Will prospectively acquire DR-CSI and sodium imaging-guided biopsies of tumor tissue in regions with different imaging characteristics. Pearson or Spearman correlations will be computed between imaging features and quantitative histological measures of cellularity, extracellular fraction, and percentages of tumor and necrosis.
Early imaging changes as predictors of clinical outcomes (Aim 2) | At baseline and 2 weeks, 3 months, and 6 months post-stereotactic radiosurgery (SRS)
  Will compute DR-CSI spectral components and TSC at each time point. Repeated measure analysis of variance will assess imaging changes over time. Will also plot trajectories of imaging biomarkers to visualize temporal patterns. Multivariate logistic regression models will evaluate early imaging changes (2 weeks and 3 months) as predictors of 6-month outcomes. Lesions will be stratified into responders (complete or partial response) and non-responders (stable disease or progression) based on their Response Assessment in Neuro-Oncology Brain Metastases assessment at 6-month post-SRS. ROC curves will assess the predictive performance of early microstructural imaging changes and the multivariate model. Primary tumor type will be included as a covariate in analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Yao, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States